CLINICAL TRIAL: NCT00660309
Title: An Open-label, Randomized, Parallel-group Study to Evaluate the Acute and Steady-state Renal Hemodynamic Responses to Aliskiren in Patients With Type 2 Diabetes Mellitus
Brief Title: A Clinical Study to Evaluate Renal Hemodynamic Responses to Aliskiren in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CSPP100A2329
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; renal disease; hypertension; renal blood flow; retinal blood flow; aliskiren; irbesartan; captopril
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Diseases; Hypertension | interventions — aliskiren; Irbesartan; Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental): On Day 1 participants received a single oral dose of 25 mg captopril. Starting on Day 2 participants received aliskiren 300 mg tablets orally once a day for 14 days.
  Interventions: Drug: Aliskiren; Drug: Captopril
- Irbesartan (Active Comparator): On Day 1 participants received a single oral dose of 25 mg captopril. Starting on Day 2 participants received irbesartan 300 mg tablets orally once a day for 14 days.
  Interventions: Drug: Irbesartan; Drug: Captopril

INTERVENTIONS:
Drug: Aliskiren — Aliskiren 300 mg tablets
  Other Names: SPP100
  Arms: Aliskiren
Drug: Irbesartan — Irbesartan 300 mg tablets
  Arms: Irbesartan
Drug: Captopril — Captopril 25 mg tablet

SUMMARY:
The study objective was to assess the effect of single and multiple doses of aliskiren on renal plasma flow, glomerular filtration rate and to compare the effects of single and multiple doses of aliskiren versus captopril or irbesartan on renal blood flow, glomerular filtration rate, and retinal blood flow in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive, male and females of non-child bearing potential patients, with type 2 diabetes mellitus (T2DM) (diagnosed at least 8 weeks before Screening), with or without renal impairment; estimated glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73 m^2, documented at least 3 months before the study start, aged 18-75 years with a minimum body weight of 50 kg and having an appropriate intravenous access as determined by the study staff, able to communicate well were enrolled in the study.
* Patients must be on a stable dose of hypoglycemic medications for at least 8 weeks prior to the study.
* Patients must be medically able to discontinue anti- hypertensive medications for the duration of the study.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus or uncontrolled T2DM (HbA1C> 11%), eGFR <40 mL/min/1.73 m^2 (calculated by the Modification of Diet in Renal Disease (MDRD) formula), renal disease not caused by diabetes or hypertension, serum potassium < 3.5 or > 5.1 mEq/L, heart failure (New York Heart Association (NYHA) Class II-IV) or history of acute/decompensated heart failure within the 6 months prior to dosing, history of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any percutaneous coronary intervention (PCI) during the 6 months prior to the baseline visit, history of malignancy including leukemia and lymphoma within past five years, hypertensive encephalopathy any time in the past or cerebrovascular accident within the 6 months prior to the baseline visit, or with history of drug or alcohol abuse within the 12 months prior to dosing were excluded from the study.
* Patients with glaucoma, or prior ocular surgery.
* Patients with renal disease not caused by diabetes or hypertension.
* Patients with history of clinically significant drug or atopic allergy, acute or chronic respiratory disease, history of malignancy, or history of myocardial infarction, unstable angina pectoris, coronary bypass surgery, or any coronary intervention (percutaneous coronary intervention; PCI) during the 6 months prior to the study.
* Patients who had used any prescription drugs which may affect the renin-angiotensin-aldosterone system or with known effect on renal hemodynamics within 2 weeks prior to dosing and during the study, over-the-counter (OTC) medication within two (2) weeks prior to dosing,
* Any surgical or medical condition which may jeopardize the patient in case of participation in the study.
* Participation in any clinical investigation within 4 weeks prior to the study.
* Donation or loss of 400 mL or more of blood within 8 weeks prior to the study.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (1):
- Novartis Investigator Site, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hollenberg NK, Fisher ND, Nussberger J, Moukarbel GV, Barkoudah E, Danser AH. Renal responses to three types of renin-angiotensin system blockers in patients with diabetes mellitus on a high-salt diet: a need for higher doses in diabetic patients? J Hypertens. 2011 Dec;29(12):2454-61. doi: 10.1097/HJH.0b013e32834c627a. PMID 22002336

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren | Irbesartan
Started | 23 (Represents participants who received one dose of Captopril.) | 22 (Represents participants who received one dose of Captopril.)
Treated With Aliskiren or Irbesartan | 22 | 21
Pharmacodynamic Analysis Set | 22 | 20
Completed | 21 | 19
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Irbesartan | Total
Number analyzed (Participants) | 23 | 22 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 56.5 (11.20) | 57.7 (8.14) | 57.1 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 17 | 12 | 29

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Renal Plasma Flow (RPF) After a Single Dose of Captopril
Description: Renal plasma flow (RPF) was measured by the clearance of para-aminohippurate (PAH) by autoanalyzer methods.
  The measure of the single dose effect (SDE) for captopril was calculated as Day 1 peak - Day 1 baseline RPF. Baseline RPF was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak RPF was obtained using a moving average concept.
Time Frame: Day 1: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and 1, 2, 3, 4 and 5 hours post-dose.
Population: Pharmacodynamics (PD) analysis set consisted of all patients with available PD data and no major protocol deviations with impact on PD data.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
mL/min/1.73m^2 | 43.32 (42.78) | 40.13 (31.70)

2. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) After a Single Dose of Captopril
Description: Glomerular filtration rate (GFR) was measured by the clearance of inulin by autoanalyzer methods.
  The measure of the single dose effect (SDE) for captopril was calculated as Day 1 peak - Day 1 baseline GFR. Baseline GFR was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak GFR was obtained using a moving average concept.
Time Frame: Day 1: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and 1, 2, 3, 4 and 5 hours post-dose.
Population: Pharmacodynamics (PD) analysis set consisted of all patients with available PD data and no major protocol deviations with impact on PD data. Analysis includes patients for whom data were available.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 16
mL/min/1.73m^2 | 11.29 (15.33) | 7.41 (12.39)

3. Primary Outcome: Change From Baseline in Renal Plasma Flow (RPF) After a Single Dose of Aliskiren or Irbesartan
Description: Renal plasma flow (RPF) was measured by the clearance of para-aminohippurate (PAH) by autoanalyzer methods.
  The measure of the single dose effect (SDE) for aliskiren and irbesartan was calculated as Day 2 peak - Day 2 baseline RPF. Baseline RPF was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak RPF was obtained using a moving average concept.
Time Frame: Day 2: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
mL/min/1.73m^2 | 37.18 (36.19) | 35.88 (35.53)

4. Primary Outcome: Change From Baseline to Steady State Trough in Renal Plasma Flow (RPF) After Aliskiren or Irbesartan
Description: Renal plasma flow (RPF) was measured by the clearance of para-aminohippurate (PAH) by autoanalyzer methods.
  This multiple dose effect at steady state (MDE_SS) was calculated as Day 15 baseline - Day 2 baseline. Baseline RPF was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values.
Time Frame: Day 2 and Day 15 at Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) .
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 18
mL/min/1.73m^2 | -5.67 (49.10) | -13.08 (27.01)

5. Primary Outcome: Change From Baseline to Steady State Peak in Renal Plasma Flow (RPF) After Aliskiren or Irbesartan
Description: Renal plasma flow (RPF) was measured by the clearance of para-aminohippurate (PAH) by autoanalyzer methods.
  This maximum multiple dose effect (MDE_Max) was calculated as Day 15 peak - Day 2 baseline. Baseline RPF was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak RPF was obtained using a moving average concept.
Time Frame: Day 2: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and Day 15: 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 18
mL/min/1.73m^2 | 24.62 (52.93) | 24.22 (38.23)

6. Primary Outcome: Change From Single Dose Peak to Steady State Peak in Renal Plasma Flow (RPF) After Aliskiren or Irbesartan
Description: Renal plasma flow (RPF) was measured by the clearance of para-aminohippurate (PAH) by autoanalyzer methods.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) was calculated as Day 15 peak - Day 2 peak. Peak RPF was obtained using a moving average concept.
Time Frame: Day 2 and Day 15: 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 18
mL/min/1.73m^2 | -12.74 (37.05) | -14.67 (35.75)

7. Secondary Outcome: Change From Baseline in Glomerular Filtration Rate (GFR) After a Single Dose of Aliskiren or Irbesartan
Description: Glomerular filtration rate (GFR) was measured by the clearance of inulin by autoanalyzer methods.
  The measure of the single dose effect (SDE) for aliskiren and irbesartan was calculated as Day 2 peak - Day 2 baseline GFR. Baseline GFR was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak GFR was obtained using a moving average concept.
Time Frame: Day 2: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 16
mL/min/1.73m^2 | 10.52 (11.22) | 10.16 (10.10)

8. Secondary Outcome: Change From Baseline to Steady State Trough in Glomerular Filtration Rate (GFR) After Aliskiren or Irbesartan
Description: Glomerular filtration rate (GFR) was measured by the clearance of inulin by autoanalyzer methods.
  This multiple dose effect at steady state (MDE_SS) was calculated as Day 15 baseline - Day 2 baseline GFR. Baseline GFR was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values.
Time Frame: Day 2 and Day 15 at Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) .
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 15
mL/min/1.73m^2 | 1.05 (10.24) | -5.67 (10.00)

9. Secondary Outcome: Change From Baseline to Steady State Peak in Glomerular Filtration Rate (GFR) After Aliskiren or Irbesartan
Description: Glomerular filtration rate (GFR) was measured by the clearance of inulin by autoanalyzer methods.
  This maximum multiple dose effect (MDE_Max) was calculated as Day 15 peak - Day 2 baseline GFR. Baseline GFR was determined as the median of the -10 minute, -5 minute predose and predose (0 hour) values. Peak GFR was obtained using a moving average concept.
Time Frame: Day 2: Baseline (10 minutes and 5 minutes pre-treatment and 0 hours) and Day 15: 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 14
mL/min/1.73m^2 | 8.69 (9.61) | 2.96 (6.98)

10. Secondary Outcome: Change From Single Dose Peak to Steady State Peak in Glomerular Filtration Rate (GFR) After Aliskiren or Irbesartan
Description: Glomerular filtration rate (GFR) was measured by the clearance of inulin by autoanalyzer methods.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) was calculated as Day 15 peak - Day 2 peak GFR. Peak GFR was obtained using a moving average concept.
Time Frame: Day 2 and Day 15: 1, 2, 3, 4 and 5 hours post-dose.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 21 | 14
mL/min/1.73m^2 | -1.71 (9.38) | -8.68 (7.05)

11. Secondary Outcome: Change in Plasma Renin Concentration (PRC) After Captopril, Aliskiren or Irbesartan
Description: The following plasma renin concentration effects were assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 Baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 Baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 Baseline / Day 2 Baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 Baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose (Baseline) and 5 hours post dose on Days 1, 2 and 15.
Population: PD analysis set. The number of patients with data available included in each analysis is indicated by 'N' [Aliskiren, Irbesartan].
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 20] | 1.18 [0.95 to 1.48] | 0.92 [0.77 to 1.09]
  SDE after aliskiren/irbesartan [N=22, 20] | 2.53 [2.09 to 3.06] | 1.04 [0.92 to 1.16]
  Steady State Trough Effect [N= 21, 19] | 4.41 [3.00 to 6.48] | 2.35 [1.48 to 3.73]
  Steady State Peak Effect [N=21, 19] | 4.81 [3.46 to 6.68] | 2.06 [1.36 to 3.12]
  Accumulation of Peak Effect [N= 21, 18] | 1.93 [1.34 to 2.76] | 1.91 [1.23 to 2.97]

12. Secondary Outcome: Change in Plasma Pro-renin Concentration After Captopril, Aliskiren or Irbesartan
Description: The following plasma pro-renin concentration effects were assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 Baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 Baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 Baseline / Day 2 Baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 Baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose (Baseline) and 5 hours post dose on Days 1, 2 and 15.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 20] | 0.97 [0.91 to 1.03] | 1.01 [0.97 to 1.05]
  SDE after aliskiren/irbesartan [N=22, 20] | 0.93 [0.89 to 0.98] | 0.96 [0.86 to 1.08]
  Steady State Trough Effect [N= 21, 19] | 1.07 [0.89 to 1.28] | 1.20 [0.98 to 1.47]
  Steady State Peak Effect [N=21, 19] | 1.10 [0.99 to 1.23] | 1.13 [0.90 to 1.43]
  Accumulation of Peak Effect [N= 21, 18] | 1.17 [1.05 to 1.32] | 1.18 [0.93 to 1.49]

13. Secondary Outcome: Change in Plasma Renin Activity (PRA) After Captopril, Aliskiren or Irbesartan
Description: PRA was measured by the trapping method and the following effects assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 baseline / Day 2 baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose and 5 hours post dose on Days 1, 2 and 15.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 20] | 1.47 [1.16 to 1.84] | 1.19 [0.83 to 1.69]
  SDE after aliskiren/irbesartan [N=22, 20] | 0.09 [0.05 to 0.15] | 1.30 [0.92 to 1.82]
  Steady State Trough Effect [N= 21, 19] | 0.12 [0.07 to 0.21] | 3.79 [1.77 to 8.12]
  Steady State Peak Effect [N=21, 18] | 0.07 [0.04 to 0.13] | 3.28 [1.67 to 6.46]
  Accumulation of Peak Effect [N= 21, 18] | 0.95 [0.83 to 1.09] | 2.67 [1.21 to 5.91]

14. Secondary Outcome: Change in Plasma Angiotensin I After Captopril, Aliskiren or Irbesartan
Description: The following angiotensin I effects were assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 Baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 Baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 Baseline / Day 2 Baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 Baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose (Baseline) and 5 hours post dose on Days 1, 2 and 15.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 19] | 2.20 [1.57 to 3.08] | 1.54 [1.08 to 2.20]
  SDE after aliskiren/irbesartan [N=22, 20] | 0.14 [0.09 to 0.25] | 0.83 [0.57 to 1.22]
  Steady State Trough Effect [N= 21, 19] | 0.24 [0.12 to 0.47] | 2.67 [1.20 to 5.93]
  Steady State Peak Effect [N=21, 18] | 0.14 [0.07 to 0.27] | 2.21 [0.96 to 5.05]
  Accumulation of Peak Effect [N= 21, 18] | 1.06 [0.63 to 1.80] | 2.71 [1.37 to 5.36]

15. Secondary Outcome: Change in Plasma Angiotensin II After Captopril, Aliskiren or Irbesartan
Description: The following angiotensin II effects were assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 Baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 Baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 Baseline / Day 2 Baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 Baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose (Baseline) and 5 hours post dose on Days 1, 2 and 15.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 19] | 0.31 [0.20 to 0.47] | 0.34 [0.22 to 0.54]
  SDE after aliskiren/irbesartan [N=22, 20] | 0.26 [0.17 to 0.38] | 1.23 [0.72 to 2.11]
  Steady State Trough Effect [N= 21, 19] | 0.43 [0.28 to 0.67] | 4.05 [1.77 to 9.26]
  Steady State Peak Effect [N=21, 18] | 0.17 [0.10 to 0.28] | 3.05 [1.39 to 6.69]
  Accumulation of Peak Effect [N= 21, 18] | 0.69 [0.43 to 1.12] | 2.49 [1.16 to 5.32]

16. Secondary Outcome: Change in Serum Aldosterone After Captopril, Aliskiren or Irbesartan
Description: The following serum aldosterone effects were assessed:
  The single dose effect (SDE) for captopril, expressed as the ratio to pre-dose measurement on Day 1, = Day 1, 5 hour / Day 1 Baseline.
  SDE for aliskiren and irbesartan = Day 2, 5 hour / Day 2 Baseline.
  Steady state trough effect (multiple dose effect at steady state; MDE_SS) = Day 15 Baseline / Day 2 Baseline.
  Steady State peak effect (maximum multiple dose effect; MDE_Max) = Day 15, 5 hour / Day 2 Baseline.
  Accumulation of peak effect from single dose to multiple dose (MDE_Acc) = Day 15, 5 hour / Day 2, 5 hour.
Time Frame: Predose (Baseline) and 5 hours post dose on Days 1, 2 and 15.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 22 | 20
ratio
  SDE after captopril [N=22, 20] | 0.58 [0.44 to 0.76] | 0.75 [0.53 to 1.05]
  SDE after aliskiren/irbesartan [N=22, 20] | 0.66 [0.49 to 0.87] | 0.65 [0.49 to 0.87]
  Steady State Trough Effect [N= 21, 19] | 0.81 [0.59 to 1.11] | 0.82 [0.61 to 1.10]
  Steady State Peak Effect [N= 21, 18] | 0.60 [0.45 to 0.79] | 0.64 [0.44 to 0.92]
  Accumulation of Peak Effect [N= 21, 18] | 0.93 [0.75 to 1.15] | 1.02 [0.81 to 1.30]

17. Secondary Outcome: Change From Baseline in Retinal Blood Flow After Aliskiren or Irbesartan
Description: Retinal blood flow was assessed using the laser Doppler technique. The blood flow in the superior temporal retinal artery in one of the eyes of each study participant was determined.
  The Single dose effect of aliskiren or irbesartan was measured as the change/difference between Day 2 and baseline measurements.
  The Multiple dose effect of aliskiren or irbesartan wsas measured as the change/difference between Day 15 and Day 2 measurements
Time Frame: Baseline (Day 1), Day 2 and Day 15.
Population: PD analysis set. This assessment was only conducted at sites with available Canon Laser Blood Flowmeter. The number of patients with data available included in each analysis is indicated by 'N' [Aliskiren, Irbesartan].
Measure: Mean (Standard Deviation); unit: µL/min
Arm/Group | Aliskiren | Irbesartan
Number analyzed (Participants) | 13 | 13
µL/min
  Single dose effect [N=13, 13] | -0.32 (1.37) | 0.43 (2.32)
  Multiple dose effect [N=13, 11] | 0.29 (1.46) | 0.35 (2.18)

ADVERSE EVENTS:
Time Frame: Study duration (14 days) and 30-days follow-up period.
Description: All patients that received at least one dose of study drug were included in the safety analysis set.
Groups:
- Captopril 25 mg: On Day 1 participants received a single oral dose of 25 mg captopril.
- Aliskiren 300 mg: Starting on Day 2 participants received aliskiren 300 mg tablets orally once a day for 14 days.
- Irbesartan 300 mg: Starting on Day 2 participants received irbesartan 300 mg tablets orally once a day for 14 days.
Arm/Group | Captopril 25 mg | Aliskiren 300 mg | Irbesartan 300 mg
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 2/45 | 5/22 | 5/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Captopril 25 mg (N=45) | Aliskiren 300 mg (N=22) | Irbesartan 300 mg (N=21)
CHEST PAIN (General disorders) | 0 | 0 | 2
BLOOD PRESSURE INCREASED (Investigations) | 0 | 2 | 0
DIZZINESS (Nervous system disorders) | 0 | 2 | 0
HEADACHE (Nervous system disorders) | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.